CLINICAL TRIAL: NCT04742777
Title: Effect of mTOR Inhibition and Other Metabolism Modulating Interventions on the Elderly: Immune, Cognitive, and Functional Consequences ((Substudy E - RAPA cMRI With LGE)
Brief Title: Effect of mTOR Inhibition & Other Metabolism Modulating Interventions on the Elderly [SubStudy Rapa & cMRI to Evaluate Cardiac Function]
Acronym: mTOR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: The Claude D. Pepper Older Americans Independence Centers (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HSC20120304H (Addendum); 5P30AG044271-07 (NIH)
Record Dates: First submitted 2021-02-01; First posted 2021-02-08 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Aging
Keywords: geriatrics
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Rapamycin 1mg for 8 weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Rapamycin (Experimental): Rapamycin 1mg for 8 weeks
  Interventions: Drug: rapamycin

INTERVENTIONS:
Drug: rapamycin — Taken orally 1mg daily for 8 weeks
  Other Names: Sirolimus

SUMMARY:
The ability to mount an effective immune response declines with age, leaving the elderly increasingly susceptible to infectious diseases and cancer. Rapamycin, an FDA approved drug to prevent transplant rejection, increases the lifespan and healthspan of mice and ameliorates age-related declines in immune responsiveness, cancer survival, and cognition in laboratory animals. Investigators are conducting a translational trial to test whether rapamycin also improves life functions in humans focusing on elderly persons (aged 70-95).

Substudy E will evaluate the Rapamycin and Cardiac Function.

DETAILED DESCRIPTION:
The main study has completed and results are reported (NCT02874924)

Purpose of Sub-study E - Rapamycin and cMRI to evaluate cardiac function:

The over-arching hypothesis is that RAPA treatment will effect simultaneous improvement in parameters known to be negatively impacted by aging. For example, systemic inflammation is higher in older individuals and contributes to the development of age-related pathologies affecting both the heart and the vasculature. In particular, evidence indicates that aging-associated alterations in inflammatory and pro-fibrotic pathways are critically involved in the etiology of age-related declines. The study team hypothesize that mTOR antagonism with RAPA will improve detrimental age-related pathologies affecting the heart in elderly humans.

ELIGIBILITY:
Inclusion Criteria:

* men and women 70-95 years of age.
* Subjects will be in good general health with all chronic diseases (hypertension, coronary artery disease, etc.) clinically stable. Selected subjects will be in good health (Per the World Health Organization good health will be defined as complete physical, mental, and social well-being and not merely the absence of disease or infirmity.
* For our purposes all diseases or infirmities will be clinically stable whether managed by medications or not.
* All ethnicities will be included.
* For cardiac and brain imaging by MRI, a pre-MRI screening questionnaire will be used to assess MRI safety and neurological health.

Exclusion Criteria:

* Diabetes, (with A1c ≥6.5 or if treated with medication affecting glucose homeostasis History of skin ulcers or poor wound healing,
* Smoking,
* Liver disease,
* Anti-coagulation,
* Treatment with drugs known to affect cytochrome P450 3A (diltiazem, erythromycin, etc) due to its role in RAPA metabolism,
* Treatment (>30days of therapy or long term) with a systemic immunosuppressant (prednisone, etc.) within the last year,
* History of recent (within 6 months) Myocardial Infarction or active Coronary Disease,
* Patients with history of recent (within 6 months) intestinal disorders,
* Exclusion criteria for MRI scan: known claustrophobia, metal implants in soft tissue of the body including pacemakers, aneurysm clips, ferrous metal fragments not anchored to bone (bullets, BBs, shrapnel, metal shavings), implanted medication pumps, and oral-facial metal appliances that are permanently secured but may result in low image quality. Participants may also be excluded for history of severe head trauma, brain injury, brain surgery, inflammation of the brain, or history of seizures.
* Positive COVID19 test.

Ages: 70 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Systolic Function | Baseline to 8 weeks
  Test whether RAPA improves systolic function in elderly subjects. Cardiac MRI will be measured before and after 8 weeks of RAPA administration using 3T MRI. From collected MRI data, the study team will quantify change in systolic volumes.
Diastolic Function | Baseline to 8 weeks
  Test whether RAPA improves diastolic function in elderly subjects.Cardiac MRI will be measured before and after 8 weeks of RAPA administration using 3T MRI. From collected MRI data, the study team will quantify change in diastolic volumes.
Aortic Cross-Sectional Area | Baseline to 8 weeks
  Test whether RAPA increases aortic compliance in elderly subjects. Aortic MRI will be measured before and after 8 weeks of RAPA using 3T MRI. The study team will quantify distal descending aortic cross-sectional area to assess aortic function/compliance effects.
Aortic Distensibility | Baseline to 8 weeks
  Test whether RAPA increases aortic compliance in elderly subjects. Aortic MRI will be measured before and after 8 weeks of RAPA using 3T MRI. The study team will quantify change in distal descending aortic distensibility to assess aortic function/compliance effects.

CONTACTS AND LOCATIONS:
Overall Officials: Dean L Kellogg, Jr., MD PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (2):
- United States (2):
  - Audie L. Murphy Memorial Veterans Hospital, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available at study completion at the time of journal publication.